CLINICAL TRIAL: NCT01808300
Title: A Randomized,Open-label,Six-sequence,Three-period,Three-treatment,Multiple Dosing Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between Pregabalin and Thioctic Acid After Oral Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug Interaction Between Pregabalin and Thioctic Acid.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unimed Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: UMPT-1; H-1212-030-449 (Registry Identifier: H-1212-030-449)
Record Dates: First submitted 2013-03-03; First posted 2013-03-11 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
MeSH Terms: interventions — Pregabalin; Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A-B-C (Experimental): Drug will be administered to according to A-B-C sequence for 3 period.
  Interventions: Drug: Pregabalin 300mg, Thioctic acid 600mg
- A-C-B (Experimental): Drug will be administered to according to A-C-B sequence for 3 period.
  Interventions: Drug: Pregabalin 300mg, Thioctic acid 600mg
- B-C-A (Experimental): Drug will be administered to according to B-C-A sequence for 3 period.
  Interventions: Drug: Pregabalin 300mg, Thioctic acid 600mg
- B-A-C (Experimental): Drug will be administered to according to B-A-C sequence for 3 period.
  Interventions: Drug: Pregabalin 300mg, Thioctic acid 600mg
- C-A-B (Experimental): Drug will be administered to according to C-A-B sequence for 3 period.
  Interventions: Drug: Pregabalin 300mg, Thioctic acid 600mg
- C-B-A (Experimental): Drug will be administered to according to C-B-A sequence for 3 period.
  Interventions: Drug: Pregabalin 300mg, Thioctic acid 600mg

INTERVENTIONS:
Drug: Pregabalin 300mg, Thioctic acid 600mg — * A: Pregabalin - Pregabalin 300mg will be administered orally twice a day for 3 days
  * B: Thioctic acid - Thioctic acid 600mg will be administered orally once a day for 3 days
  * C: Pregabalin plus Thioctic acid - Pregabalin plus Thioctic acid same way as A and B

SUMMARY:
A randomized, open-label, six-sequence, three-period, three-treatment, multiple dosing clinical trial to investigate the pharmacokinetic drug interaction between Pregabalin and Thioctic acid after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight ae least 50kg and BMI(body mass index) within the range of 18 to 27kg/m2
2. Provision of signed written informed consent
3. Acceptable physical examination and clinical examination, during screening

Exclusion Criteria:

1. A subject with clinical evidence or history of hepatic (including carrier of hepatitis virus), renal, respiratory, endocrine, neurologic, immunologic, hematologic, oncologic, psychiatric, or cardiovascular disease
2. A subject with a history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
3. A subject with history of allergies including study drug (pregabalin or thioctic acid) or other drug allergies (aspirin, antibiotics, etc.), or history of clinically significant allergies
4. A subject whose lab test results are as follows: AST(SGOT), ALT(SGPT) > 1.5 x upper limit of reference range
5. Presence or history of drug abuse or positive result in urine drug screening test
6. Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
7. Participation in clinical trials of any drug within 60 days prior to the participation of the study
8. Blood donation during 2 months or apheresis during 1 month before the study
9. Use of alcohol over 21 units/weeks
10. Smoker who smoke more than 10 cigarettes per day or who cannot stop smoking during the study period (from 24 hours before hospitalization to discharge)
11. Use of caffeine drink during the study period(from 24 hours before hospitalization to discharge)
12. A subject who takes grapefruit, grapefruit juice, or grapefruit-containing products during the study
13. Judged to be inappropriate for the study by the investigator after reviewing clinical laboratory results or other reasons.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss / Cmax of pregabalin and thioctic acid | 2d (9d, 16d): 0h (predose:Thioctic acid), 12h (pre-dose:Pregabalin), 3d(10d, 17d): 0h (pre-dose), 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12h, 24h

SECONDARY OUTCOMES:
Ctrough,ss / Tmax,ss / t½ / CL/F of pregabalin and thioctic acid | 2d (9d, 16d): 0h (predose:Thioctic acid), 12h (pre-dose:Pregabalin), 3d(10d, 17d): 0h (pre-dose), 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12h, 24h

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Derived] Rhee SJ, Lee H, Ahn LY, Lim KS, Yu KS. Lack of a Clinically Significant Pharmacokinetic Interaction Between Pregabalin and Thioctic Acid in Healthy Volunteers. Clin Ther. 2018 Oct;40(10):1720-1728.e2. doi: 10.1016/j.clinthera.2018.08.016. Epub 2018 Sep 18. PMID 30241687